CLINICAL TRIAL: NCT02457780
Title: Mind-Body Treatment for WTC Responders With Comorbid PTSD and Respiratory Illness
Brief Title: Stress Management Program for World Trade Center (WTC) Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01OH010524-01 (NIH)
Record Dates: First submitted 2015-05-04; First posted 2015-05-29 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: PTSD; Signs and Symptoms, Respiratory
Keywords: PTSD; Trauma; World Trade Center; Respiratory; Mind-Body
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Signs and Symptoms, Respiratory; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation Response Resiliency Program (Experimental): The Relaxation Response Resiliency Program (3RP) is an 8-session (90min/session) group based intervention which includes a variety of skills and techniques designed to address chronic stress. Techniques used include psychoeducation on healthy lifestyle behaviors, goal-setting, CBT skills, relaxation training and self-monitoring.
  Interventions: Behavioral: Relaxation Response Resiliency Program (3RP)
- Health Enhancement Program (Active Comparator): The Health Enhancement Program (HEP) is an 8-session (90min/session) group based intervention which includes psychoeducation and self-monitoring of health behaviors (e.g., sleep hygiene, nutrition, exercise, substance use etc).
  Interventions: Behavioral: Health Enhancement Program (HEP)

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program (3RP) — The 3RP is designed to decrease psychiatric and physical health symptoms and build resiliency by teaching skills to (1) elicit the relaxation response, (2) decrease stress reactivity and (3) increase social connectedness. Eliciting the relaxation response involves sustained mental focus with an attitude of receptive awareness with strategies aimed at reducing muscle tension, breathing rate, heart rate, and blood pressure. Decreasing stress reactivity involves increasing awareness of the stress response and learning skills to proactively address stress. Increasing connectedness involves skills to promote positive growth, self-efficacy and social support. Other skills and experiential exercises focus on increasing acceptance, optimism, empathy, and appreciation to promote resiliency.
  Other Names: Stress Management and Resiliency Training (SMART)
  Arms: Relaxation Response Resiliency Program
Behavioral: Health Enhancement Program (HEP) — The HEP is designed to address comorbid physical and mental health symptoms via psychoeducation, self-monitoring and goal setting techniques. It is an 8 session manualized group intervention which addresses topics including sleep hygiene, nutrition, exercise, working with a healthcare team, and substance use. The program uses a variety of in-session activities to engage participants in discussion related to self-care and wellness principles. Relapse prevention and long-term goal setting are addressed. The program is designed to be implemented by professionals with a background in mental health.
  Arms: Health Enhancement Program

SUMMARY:
Many responders to the World Trade Center (WTC) disaster continue to experience significant mental and physical health problems. Two of the most common health problems, post-traumatic stress disorder (PTSD) symptoms and respiratory illness, often occur together. Mental health conditions, such as PTSD, make physical illnesses worse and interfere with treatment. The primary goal of this study is to test a mind-body treatment designed to reduce both PTSD and respiratory symptoms.

DETAILED DESCRIPTION:
Mind-body interventions including relaxation training and other coping skills are effective for patients with both mental and physical health problems. A leading mind-body treatment is the Relaxation Response Resiliency Program (3RP) developed at Harvard. This treatment has been shown to reduce both mental and physical health symptoms.

The objective of this study is to adapt the 3RP to WTC responders and test its ability to reduce both PTSD and respiratory symptoms. This treatment will be compared to a Health Enhancement Program that addresses negative health behaviors. The investigators will randomly assign 175 patients with ongoing WTC-related PTSD and respiratory illness to the 3RP or Health Enhancement Program and will assess outcomes immediately after the treatment and at 3 and 6 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* PCL score equal to or greater than 35
* 2 or more lower respiratory symptoms

Exclusion Criteria:

* Regular elicitation of the relaxation response
* History of psychosis
* Current unmanaged bipolar disorder
* History of suicide attempt --OR-- current ideation with plan or intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-report WTC-related PTSD Symptoms | Change from baseline in WTC-related PTSD symptoms at 6-months
  Assessed via self-report (PTSD Checklist Specific Stressor; PCL-S)
Clinician Rated WTC-related PTSD Symptoms | Change from baseline in WTC-related PTSD symptoms at 6-months
  Assessed via clinician interview (SCID for DSM-IV-TR).

SECONDARY OUTCOMES:
Lower Respiratory Symptoms | Change from baseline in lower respiratory symptoms at 6-months
  Assessed via self-report
Pulmonary Functioning | Change from baseline in pulmonary functioning at 6-months
  Assessed via spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gonzalez, PhD, Principal Investigator — Stony Brook University Department of Psychiatry
Locations (1):
- Stony Brook University, Putnam Hall, Stony Brook, New York, United States